CLINICAL TRIAL: NCT07389837
Title: Dose-Response Effects of Maple Syrup Carbohydrate Ingestion (60, 90, 120 g/h) on 20-km Cycling Time-Trial Performance, Substrate Oxidation, and Perceptual Responses in Trained Male Cyclists
Brief Title: Maple Syrup Carbohydrate Dose-Response on 20-km Cycling Time-Trial Performance
Acronym: MAPLE-DR
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Montréal (Other)
Collaborators: Natural Sciences and Engineering Research Council, Canada (Other); Montreal Heart Institute (Other); Mitacs (Industry); Quebec Maple Syrup Producers (Unknown); Quebec Cycling Federation (Unknown)
Responsible Party: Principal Investigator, Jonathan Tremblay, Full Professor, Université de Montréal
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ICM 2026-3568
Record Dates: First submitted 2026-01-02; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Exercise; Endurance Cycling Performance; Carbohydrate Intolerance; Sport Nutrition
Keywords: 13C-glucose; cycling exercise; endurance performance; carbohydrate; substrate oxidation
MeSH Terms: conditions — Motor Activity; Glucose-Galactose Malabsorption

STUDY DESIGN:
Intervention Model Description: This is a randomized, double-blind, placebo-controlled, crossover trial designed to maximize statistical power. Each participant will serve as their own control, completing four experimental conditions in computer-randomized order.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Maple syrup providing 60g of CHO per hour (Experimental): The protocol begins with a 10-minute warm-up at 100 W, followed by a 120-minute constant-load cycling phase at 65% PPO, during which the 60 g/h maple syrup solution is consumed every 15 minutes as the main intervention. Neuromuscular fatigue is assessed four times (baseline, 60 min, 120 min into the constant-load, and post-TT) using two 6-second all-out seated sprints (from a 100 W rolling start); these two sprints are separated by a 1-minute active recovery at 100 W, after which the 65% PPO cycling is immediately resumed for the in-exercise timepoints. The constant-load phase is concluded by a 5-minute complete recovery, immediately followed by the 20-km self-paced Time Trial (completed without fluids), with the final set of sprints performed immediately after the TT to assess residual fatigue.
  Interventions: Dietary Supplement: Maple Syrup Beverages; Dietary Supplement: placebo beverage; Other: Pre-Trial Meals; Procedure: D₂O Fluid Absorption; Behavioral: Time Trial Performance; Procedure: Substrate Oxidation; Procedure: Blood Metabolites; Diagnostic Test: Gastrointestinal Symptoms; Diagnostic Test: Perceptual Responses; Diagnostic Test: Neuromuscular Fatigue; Other: Hedonic Ratings; Other: Blinding Integrity
- Maple syrup providing 90g of CHO per hour (Experimental): The protocol begins with a 10-minute warm-up at 100 W, followed by a 120-minute constant-load cycling phase at 65% PPO, during which the 90 g/h maple syrup solution is consumed every 15 minutes as the main intervention. Neuromuscular fatigue is assessed four times (baseline, 60 min, 120 min into the constant-load, and post-TT) using two 6-second all-out seated sprints (from a 100 W rolling start); these two sprints are separated by a 1-minute active recovery at 100 W, after which the 65% PPO cycling is immediately resumed for the in-exercise timepoints. The constant-load phase is concluded by a 5-minute complete recovery, immediately followed by the 20-km self-paced Time Trial (completed without fluids), with the final set of sprints performed immediately after the TT to assess residual fatigue.
  Interventions: Dietary Supplement: Maple Syrup Beverages; Dietary Supplement: placebo beverage; Other: Pre-Trial Meals; Procedure: D₂O Fluid Absorption; Behavioral: Time Trial Performance; Procedure: Substrate Oxidation; Procedure: Blood Metabolites; Diagnostic Test: Gastrointestinal Symptoms; Diagnostic Test: Perceptual Responses; Diagnostic Test: Neuromuscular Fatigue; Other: Hedonic Ratings; Other: Blinding Integrity
- Maple syrup providing 120g of CHO per hour (Experimental): The protocol begins with a 10-minute warm-up at 100 W, followed by a 120-minute constant-load cycling phase at 65% PPO, during which the 120 g/h maple syrup solution is consumed every 15 minutes as the main intervention. Neuromuscular fatigue is assessed four times (baseline, 60 min, 120 min into the constant-load, and post-TT) using two 6-second all-out seated sprints (from a 100 W rolling start); these two sprints are separated by a 1-minute active recovery at 100 W, after which the 65% PPO cycling is immediately resumed for the in-exercise timepoints. The constant-load phase is concluded by a 5-minute complete recovery, immediately followed by the 20-km self-paced Time Trial (completed without fluids), with the final set of sprints performed immediately after the TT to assess residual fatigue.
  Interventions: Dietary Supplement: Maple Syrup Beverages; Dietary Supplement: placebo beverage; Other: Pre-Trial Meals; Procedure: D₂O Fluid Absorption; Behavioral: Time Trial Performance; Procedure: Substrate Oxidation; Procedure: Blood Metabolites; Diagnostic Test: Gastrointestinal Symptoms; Diagnostic Test: Perceptual Responses; Diagnostic Test: Neuromuscular Fatigue; Other: Hedonic Ratings; Other: Blinding Integrity
- Placebo (Placebo Comparator): The protocol begins with a 10-minute warm-up at 100 W, followed by a 120-minute constant-load cycling phase at 65% PPO, during which the placebo solution (sweetened water, with sotolon for maple taste) is consumed every 15 minutes as the main intervention. Neuromuscular fatigue is assessed four times (baseline, 60 min, 120 min into the constant-load, and post-TT) using two 6-second all-out seated sprints (from a 100 W rolling start); these two sprints are separated by a 1-minute active recovery at 100 W, after which the 65% PPO cycling is immediately resumed for the in-exercise timepoints. The constant-load phase is concluded by a 5-minute complete recovery, immediately followed by the 20-km self-paced Time Trial (completed without fluids), with the final set of sprints performed immediately after the TT to assess residual fatigue.
  Interventions: Dietary Supplement: Maple Syrup Beverages; Dietary Supplement: placebo beverage; Other: Pre-Trial Meals; Procedure: D₂O Fluid Absorption; Behavioral: Time Trial Performance; Procedure: Substrate Oxidation; Procedure: Blood Metabolites; Diagnostic Test: Gastrointestinal Symptoms; Diagnostic Test: Perceptual Responses; Diagnostic Test: Neuromuscular Fatigue; Other: Hedonic Ratings; Other: Blinding Integrity

INTERVENTIONS:
Dietary Supplement: Maple Syrup Beverages — Pure maple syrup is diluted in water and mixed with electrolytes (sodium, potassium, magnesium) to resemble a sports drink. Participants receive one of three carbohydrate doses (60, 90, or 120 g per hour). Drinks are ingested every 15 minutes during 120 minutes of cycling, for a total of ~750 mL per hour. All doses have the same volume, temperature, electrolyte content, and schedule.
Dietary Supplement: placebo beverage — Participants receive a calorie-free electrolyte drink designed to mimic maple syrup. Sotolon (maple aroma) and stevia are added in small amounts to reproduce sweetness, flavor, and smell without providing energy. The drink is administered in identical volumes and timing to the maple syrup beverages (~750 mL per hour, every 15 minutes).
Other: Pre-Trial Meals — To control nutrition before each trial, participants are provided with a standardized dinner the night before and a standardized breakfast 2-3 hours before testing. Meals contain the same calories and macronutrient distribution across all sessions. Participants must also replicate their training during the previous 48 hours.
Procedure: D₂O Fluid Absorption — At 30 minutes of cycling, participants ingest a small, safe dose of deuterium oxide (7-8 mL) to measure fluid absorption and gastric emptying. Additional blood samples are collected at +32, +35, and +40 minutes to capture early absorption. Urine is collected to measure deuterium enrichment and validate absorption kinetics.
Behavioral: Time Trial Performance — After 120 minutes of steady cycling, participants complete a 20-km self-paced time trial. Only distance is displayed. The primary outcome is completion time; mean power is analyzed as supportive information.
Procedure: Substrate Oxidation — Energy metabolism is measured using indirect calorimetry and ¹³C-sucrose breath enrichment. Samples are collected at rest and every 30 minutes during exercise to quantify carbohydrate and fat use, distinguishing ingested vs. stored carbohydrate oxidation. Urine and sweat correct protein oxidation.
Procedure: Blood Metabolites — Blood samples collected every 30 minutes measure glucose, insulin, lactate, and fatty acids. Samples are stored for later analysis of hormonal and metabolic responses.
Diagnostic Test: Gastrointestinal Symptoms — Participants rate stomach symptoms (0-10 scale) before exercise, every 30 minutes during cycling, and after the time trial. Scores quantify total, upper, and lower GI discomfort.
Diagnostic Test: Perceptual Responses — Effort and muscle pain are assessed using the Borg CR100 scale during exercise and throughout the time trial at preset intervals.
Diagnostic Test: Neuromuscular Fatigue — Participants perform two 6-second maximal sprints at baseline, 60 and 120 minutes of cycling, and after the time trial. Peak power, cadence, and torque assess fatigue progression and recovery.
Other: Hedonic Ratings — Immediately post-exercise, a 0-100 mm scale evaluates sweetness, flavor intensity, and overall liking to assess palatability of each drink.
Other: Blinding Integrity — Bang's Blinding Index is calculated from participant guesses of drink identity to confirm whether blinding was successful.

SUMMARY:
The goal of this clinical trial is to learn whether maple syrup can be used as a natural carbohydrate source to help trained male cyclists perform better during long-duration cycling. The study also aims to learn how different amounts of maple syrup affect energy use in the body, stomach comfort, and feelings of effort and fatigue.

The main questions the study aims to answer are:

* Does consuming more carbohydrate from maple syrup help participants finish a 20-kilometer cycling time trial faster?
* How do different amounts of maple syrup change how the body uses carbohydrates and fats during long exercise?
* Are higher amounts of maple syrup easy for participants to tolerate without stomach problems?

Researchers will compare four drinks:

1. A placebo drink (a look-alike drink with no calories),
2. A drink that provides 60 grams of carbohydrate per hour,
3. A drink that provides 90 grams per hour, and
4. A drink that provides 120 grams per hour.

They will compare these drinks to see whether higher carbohydrate amounts lead to better cycling performance and how each dose affects comfort and metabolism.

Participants will:

* Attend a screening visit that includes a health check and a glucose tolerance test.
* Complete a fitness test to measure their aerobic capacity and practice the cycling tests used in the study.
* Take part in four separate exercise sessions in random order. Each session includes:
* Drinking one of the four study beverages during 2 hours of steady cycling,
* Completing two short, all-out 6-second sprints during the ride,
* Completing a 20-kilometer cycling time trial as fast as possible,
* Reporting stomach symptoms and perceptions of effort,
* Providing breath, blood, urine, and sweat samples so researchers can measure how their body uses fuel.

All drinks will look, taste, and smell similar so participants cannot tell which one they are receiving. Meals before each session will be provided to keep conditions the same across visits.

This study may help athletes and active people choose natural carbohydrate sources that support both performance and comfort during long endurance exercise. The findings may also guide future research on the use of maple syrup as a sports nutrition option.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-45 years.
* Relative VO2max: >55 mL·min-¹·kg-¹ for level 3; >65 mL·min-¹·kg-¹ for level 4.
* Peak Power Output (PPO): >4.6 W·kg-¹ (absolute PPO >320 W).
* Training History: >5 hours/week of cycling-specific training; >1 year of consistent endurance training.
* No history of metabolic disorders, gastrointestinal issues, or contraindications to exercise testing.

Exclusion Criteria:

* Current or past metabolic disorders (diabetes, metabolic syndrome)
* Cardiovascular disease or abnormal ECG at rest
* Gastrointestinal disorders (IBS, Crohn's, celiac disease)
* Food allergies or intolerances (particularly maple, fructose)
* Current use of medications affecting metabolism
* Smoking or nicotine use
* Alcohol consumption >14 units/week
* Recent illness or injury (<4 weeks)
* Participation in other clinical trials (<3 months)
* Unable to maintain consistent training during study period

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Assess the dose-response effect of maple syrup carbohydrate ingestion (0, 60, 90, 120 g·h-¹) on 20-km cycling time-trial performance in trained male cyclists. | Immediately after completion of the 20-km time trial during each experimental visit
  20-km time trial completion time (minutes), measured at the end of each experimental visit.

SECONDARY OUTCOMES:
Substrate oxidation rates during exercise | At rest, immediately before exercise, and every 30 minutes during 120 minutes of constant-load cycling
  Exogenous and endogenous carbohydrate oxidation, fat oxidation, and protein oxidation rates (g·min-¹) measured via ¹³C stable isotope breath enrichment and indirect calorimetry.
Plasma metabolite concentrations | Measured before beverage ingestion, immediately pre-exercise, every 30 minutes during the 120-minute constant-load cycling, and immediately post-exercise (before the time trial).
  Plasma glucose, insulin, lactate, and free fatty acid concentrations sampled before beverage ingestion, pre-exercise, every 30 minutes during constant-load exercise, and immediately after.
Ratings of perceived effort during exercise | Assessed 3 minutes after exercise begins; every 30 minutes during the constant-load cycling (30, 60, 90, 120 min); and at approximately 126, 127, 130, 136, and 145 minutes (corresponding to 0.5, 5, 10, 15, and 20 km during the time trial)
  Ratings of perceived effort (CR100 scale, 0-100) collected after 3 minutes and every 30 minutes during constant-load exercise, and during the time trial.
Assess gastrointestinal tolerance and symptoms across maple syrup doses and placebo. | Measured pre-exercise; every 30 minutes during the 120-minute constant-load cycling (30, 60, 90, 120 min); and immediately after the time trial.
  Gastrointestinal distress scores (0-10 on a modified visual analog scale, mVAS), rated pre-exercise, every 30 minutes during the constant-load exercise, and post-TT; includes composite scores for total, upper, and lower GI symptoms.
Peak power output during maximal sprints | Baseline, 60 minutes, 120 minutes, and immediately after time trial
  Peak power output (watts) from two 6-second maximal sprints performed at baseline, 60 minutes, 120 minutes, and post-time trial.
Mean power output during 20-km time trial | Approximately 25-30 minutes (continuously recorded during the 20-km time trial)
  Mean power output (watts) recorded continuously during the 20-km time trial.

OTHER OUTCOMES:
Hedonic ratings for beverage sweetness, flavor, and liking | Immediately after time trial completion
  Hedonic ratings for sweetness, flavor intensity, and overall liking (0-100 mm visual analog scale) assessed immediately post-exercise.
Explore correlations between substrate oxidation rates and TT performance. | Evaluated using oxidation values measured during cycling (at rest, pre-exercise, and at 30, 60, 90, 120 min) and TT performance measured at approximately 150-155 minutes (immediately after time trial completion)
  Correlation coefficients (e.g., Pearson's r) between exogenous/endogenous oxidation rates and TT time to completion or mean power output.
Examine inter-individual variability in dose-response patterns for performance outcomes. | Calculated from repeated TT measurements collected at each of 4 experimental visits over approximately 4-6 weeks
  Within-subject and inter-individual coefficients of variation for TT time to completion and mean power output across doses.
Assess gastrointestinal absorption kinetics across maple syrup doses and placebo. | Measured via plasma samples at baseline, 30 min (pre-ingestion), and at +32, +35, +40 min, then every 30 min during cycling (60, 90, 120 min), plus within 30 minutes after time trial completion (approximately 150-180 min)
  Deuterium oxide (D2O) tracer kinetics, including absorption rate constant, time-to-peak plasma enrichment (tmax), and area under the curve (AUC), derived from plasma and urine D/H enrichment samples.
Explore whether individual characteristics (e.g., body weight, training volume) moderate the dose-response effects of maple syrup on endurance performance. | Moderation assessed using TT outcomes collected at each of 4 experimental visits over approximately 4-8 weeks, combined with participant baseline characteristics collected at screening visit
  Moderation analysis using interaction terms in linear mixed-effects models (e.g., carbohydrate dose × body weight) for TT time to completion.
Explore plasma metabolomic signatures associated with carbohydrate dose and performance. | Baseline (before beverage ingestion), immediately before exercise, at 60 minutes of constant-load cycling, pre-TT (~125 minutes after beginning constand-load cycling), and post-TT (~150-160 minutes).
  Untargeted metabolomic profiling via high-resolution liquid chromatography-tandem mass spectrometry (LC-MS/MS) on plasma samples collected at before beverage ingestion, before the start of exercise, at 60 minutes into constant-load exercise, pre- and post-TT; focuses on pathways such as glycolysis, lipid oxidation, and amino acid metabolism.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Tremblay, PhD, Principal Investigator — Université de Montréal
Locations (1):
- Centre EPIC, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified, row-level participant data collected in this trial, including: 20-km TT completion time and mean power; VO2max and PPO from incremental test; whole-body substrate oxidation (carbohydrate, fat, protein) and exogenous/endogenous carbohydrate oxidation from 13C breath enrichment; respiratory gas exchange (VO2, VCO2); plasma biomarkers (glucose, insulin, lactate, free fatty acids) at scheduled time points; D2O fluid absorption kinetics (rate constant, tmax, AUC); gastrointestinal symptom scores (mVAS); perceptual responses (Borg CR100 effort and muscle pain); neuromuscular fatigue metrics (6-s sprints: peak power, cadence, torque) at all timepoints; hedonic ratings (sweetness, flavor, overall liking); blinding guesses (Bang's index); and baseline demographics (age, body mass). Direct identifiers will be removed; dates and rare combinations will be masked per de-identification standards.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: 12 months after primary results publication and for at least 5 years
Access Criteria: Qualified researchers at accredited institutions may request access to de-identified IPD and supporting materials (protocol, SAP, and analytic code if available). Requests must include a study synopsis, analysis plan, variables needed, and documentation of IRB/ethics approval. The PI/sponsor data access committee will review for scientific merit, feasibility, and privacy protection. Approved users must sign a Data Use Agreement prohibiting re-identification, onward sharing, and commercial use; publications must acknowledge the original study. Access will be time-limited via a secure repository with role-based permissions, encryption, and audit logs; only aggregate results may be publicly released. Linkage to external datasets requires explicit approval.
URL: https://bioenergeticslab.ca/en/contact

REFERENCES:
- [Background] Cermak NM, van Loon LJ. The use of carbohydrates during exercise as an ergogenic aid. Sports Med. 2013 Nov;43(11):1139-55. doi: 10.1007/s40279-013-0079-0. PMID 23846824
- [Background] Stellingwerff T, Cox GR. Systematic review: Carbohydrate supplementation on exercise performance or capacity of varying durations. Appl Physiol Nutr Metab. 2014 Sep;39(9):998-1011. doi: 10.1139/apnm-2014-0027. Epub 2014 Mar 25. PMID 24951297
- [Background] Jeukendrup AE. Carbohydrate and exercise performance: the role of multiple transportable carbohydrates. Curr Opin Clin Nutr Metab Care. 2010 Jul;13(4):452-7. doi: 10.1097/MCO.0b013e328339de9f. PMID 20574242
- [Background] Vandenbogaerde TJ, Hopkins WG. Effects of acute carbohydrate supplementation on endurance performance: a meta-analysis. Sports Med. 2011 Sep 1;41(9):773-92. doi: 10.2165/11590520-000000000-00000. PMID 21846165
- [Background] Smith JW, Zachwieja JJ, Peronnet F, Passe DH, Massicotte D, Lavoie C, Pascoe DD. Fuel selection and cycling endurance performance with ingestion of [13C]glucose: evidence for a carbohydrate dose response. J Appl Physiol (1985). 2010 Jun;108(6):1520-9. doi: 10.1152/japplphysiol.91394.2008. Epub 2010 Mar 18. PMID 20299609
- [Background] Hearris MA, Pugh JN, Langan-Evans C, Mann SJ, Burke L, Stellingwerff T, Gonzalez JT, Morton JP. 13C-glucose-fructose labeling reveals comparable exogenous CHO oxidation during exercise when consuming 120 g/h in fluid, gel, jelly chew, or coingestion. J Appl Physiol (1985). 2022 Jun 1;132(6):1394-1406. doi: 10.1152/japplphysiol.00091.2022. Epub 2022 Apr 21. PMID 35446596
- [Background] Lavoie L, Tremblay J. Ingestion of maple-based and other carbohydrate sports drinks: effect on sensory perceptions during prolonged exercise. J Int Soc Sports Nutr. 2020 Dec 9;17(1):63. doi: 10.1186/s12970-020-00384-3. PMID 33298104
- [Background] De Pauw K, Roelands B, Cheung SS, de Geus B, Rietjens G, Meeusen R. Guidelines to classify subject groups in sport-science research. Int J Sports Physiol Perform. 2013 Mar;8(2):111-22. doi: 10.1123/ijspp.8.2.111. PMID 23428482